CLINICAL TRIAL: NCT04080817
Title: Prospective, Randomized, Clinical & Experimental Controlled Noninvasive Study for Neolexon® Aphasia-App in Acute Aphasia After Stroke
Brief Title: Neolexon® Aphasia-App in Acute Aphasia After Stroke
Acronym: Lexi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Lars Kellert, Principal Investigator, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-068
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Aphasia, Acquired; Stroke, Acute
Keywords: Stroke; Aphasia; Speech therapy; Computer based
MeSH Terms: conditions — Aphasia; Stroke; Communication Disorders | interventions — Speech Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neolexon Therapy (Experimental)
  Interventions: Device: Neolexon; Other: Self training
- Standard logopedic therapy (Active Comparator)
  Interventions: Other: Speech therapy; Other: Self training

INTERVENTIONS:
Device: Neolexon — Application (Neolexon) on Tablet. Same frequency & intensity as in the other interventions
  Arms: Neolexon Therapy
Other: Speech therapy — standard logopedic speech therapy. Same frequency & intensity as in the other interventions
  Arms: Standard logopedic therapy
Other: Self training — Same frequency & intensity as in the other interventions

SUMMARY:
Up to now there is proven evidence of traditional logopedic therapy in aphasia, but recent computer-based algorithms also showed their evidence so far. Due to small and heterogenous study populations further trials are urgently needed. This prospective, randomized, clinical & experimental controlled noninvasive study is intended to provide data for the therapy of an individual approach in aphasia patients.

DETAILED DESCRIPTION:
The prospective, randomized, clinical & experimental controlled noninvasive study (Lexi) is intended to start in 10/2019. Adult and German speaking patients suffering from aphasia after stroke who give informed consent and whose life expectancy is estimated above 1 year are included and will be followed up for 3 months. If informed consent is not available their legal guardian will have to provide written informed consent for their contribution.

After Randomization participants are divided into two different groups:

Patients receiving a standard logopedic speech treatment versus individuals working with a computer-based solution (Neolexon® App on mobile devices). Both groups will also have self-training and therefore frequency and intensity of this is also going to be analyzed as well as in the clinical surrounding.

There will be three different major ward rounds in both groups during the trial period where scales scoring the severity of aphasia are collected and compared (i.e. AABT or LAST).

Furthermore epidemiologic data and stroke scales (i.e. NIHSS, mRS) are evaluated. The last round will be the follow-up after 3 months. Lexi will provide new data to fill the gap of organizational barriers and structural problems. Our aim is to show modern alternative therapy algorithms that approach the individual problem to offer a potential tailored solution to patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Acute Aphasia after stroke (ischemic oder hemorrhagic)
* Life expectancy ≥ 1 year
* Informed consent (presumed)
* Mother tongue: german

Exclusion Criteria:

* Age < 18 years
* Missing aphasia
* Life expectancy < 1 year
* Mother tongue: other then german

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Epidemiologic Data | 3 months
  age, etiology of stroke, symptoms of stroke, specific stroke therapy (i.e. intravenous thrombolysis/recanalisation),
NIHSS | 3 months
  NIHSS "National Institutes of Health Stroke Scale". It is a Scoring System , which objectively quantifies severity of stroke based on weighted evaluation findings.
  Scoring: https://www.stroke.nih.gov/documents/NIH_Stroke_Scale.pdf Calculating/Interpreting: Higher Scores predict poor outcome and high severity of stroke. Low Scores are associated with minimal mortality and good prognosis. The minimum score being 0, and the maximum score being 42. Subscales are summed to a total Score (high score means worse prognosis, low score indicates a good prognosis.
p-mRS | 3 months
  premorbid Modified Rankin Scale (mRS): It is a Scoring System , which objectively quantifies disability before stroke in daily activities. Same questions/scores as in "Outcome 4".
mRS | 3 months
  1. Modified Rankin Scale (mRS): It is a Scoring System , which objectively quantifies disability after stroke in daily activities.
  2. Scoring http://www.strokecenter.org/wp-content/uploads/2011/08/modified_rankin.pdf
  3. There is only one total score. The minimum possible score is 0 and the maximum possible score is 6. A high score means worse prognosis/dead, low score indicates a good prognosis.
  4. It is summed.
BI | 3 months
  Barthel Index
LAST | 3 months
  Language Screening Test
AABT | 3 months
  Aachener Aphasie Bedside Test
ACL | 3 months
  Aphasie Check Liste

SECONDARY OUTCOMES:
EQ-5D-5L | 3 months
  "US 5-level EuroQol 5-dimensional questionnaire" Its a scoring tool, which objectively quantfies life quality. It consists of two seperate parts.
  2. I: Scoring the Descriptive System with five dimensions. Each dimension has 5 boxes. 1-5 are scored as 1-5.
  -> There should be only 1 response for each dimension, Missing values can be coded as '9'. Ambiguous values should be treated as missing values.
  Each health state is referred to in terms of a 5 digit code 11111 (best health state), 55555 (worst health state)
  II: Scoring the VAS (visual analogue scale): This scale is numbered from 0 to 100. (100 means the best health you can imagine. 0 means the worst health you can imagine.) An X should be marked in the scale and then the number into a box. (Missing values should be coded as '999'.) https://euroqol.org/docs/Sample_UK__English__EQ-5D-5L_Paper_Self_complete.pdf, https://apersu.ca/wp-content/uploads/2017/07/Measuring-and-valuing-health-using-the-EQ-5D.pdf
BDI | 3 months
  Beck Depression Inventory. A self-scoring tool to objectively count the severity of depressive symptoms consisting of 21 questions. Each question ranges from 0 to 3 points. Subscales are summed. Maximum score is possible at 63 (21x3) and minimal score being 0."
  Levels of Depression 1-10 These ups and downs are considered normal 11-16 Mild mood disturbance 17-20 Borderline clinical depression 21-30 Moderate depression 31-40 Severe depression Over 40 Extreme depression"
  Source:
  https://www.google.com/url?sa=t&rct=j&q=&esrc=s&source=web&cd=2&ved=2ahUKEwjd3u362rvkAhVSZ1AKHZJ4CCAQFjABegQIABAC&url=https%3A%2F%2Fwww.enhertsccg.nhs.uk%2Fsites%2Fdefault%2Ffiles%2Fpathways%2FBeck%2527s%2520Depression%2520Inventory_0.docx&usg=AOvVaw3MwAYfr0zL21nK88Cn4VTG"

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Feil, MD, Principal Investigator — Ludwig Maximlians University (LMU) Munich
Locations (1):
- Ludwig Maximilians University (LMU) Munich, Department of Neurology with Friedrich-Baur Institute, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wischmann J, Brasch L, Franzen J, Schwierz J, Kovalenko O, Gutmann A, Erbert F, Bussmann L, Lauer J, Dumberger C, Mandl A, Mehringer M, Munsterer A, Spitzer J, Winterhalter L, Frank V, Rheinwald M, Lehner K, Ammer F, Pfahler A, Lampart S, Young C, Young P, Goettert B, Bitzan M, Rinder S, Meier O, Feil K, Kellert L. Tablet-Assisted Speech and Language Therapy for Acute Post-Stroke Aphasia: A Randomized Clinical Trial (LEXI Study). Eur J Neurol. 2025 Dec;32(12):e70443. doi: 10.1111/ene.70443. PMID 41294376
- [Derived] Thunstedt DC, Young P, Kupper C, Muller K, Becker R, Erbert F, Lehner K, Rheinwald M, Pfahler A, Dieterich M, Kellert L, Feil K. Follow-Up in Aphasia Caused by Acute Stroke in a Prospective, Randomized, Clinical, and Experimental Controlled Noninvasive Study With an iPad-Based App (Neolexon(R)): Study Protocol of the Lexi Study. Front Neurol. 2020 Apr 30;11:294. doi: 10.3389/fneur.2020.00294. eCollection 2020. PMID 32425873